CLINICAL TRIAL: NCT06775626
Title: Changes in Body Composition and Sport Performance Among Young Female Soccer Players Using Subdermic Etonogestrel (Implanon NXT)
Brief Title: Body Composition and Sport Performance Among Young Female Soccer Players Using Subdermic Etonogestrel
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was suspended due to non-compliance with the partnership agreement between the research team and the company that would supply Implanon. Therefore, it was not possible to continue the study
Sponsor: Maíta Poli de Araújo (Other)
Collaborators: Organon (Industry)
Responsible Party: Sponsor-Investigator, Maíta Poli de Araújo, Assistant professor in the Department of Gynecology at Federal University of São Paulo, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 76907423.1.0000.5505
Record Dates: First submitted 2024-12-27; First posted 2025-01-15 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Menstrual Symptoms
Keywords: menstrual symptoms; etonogestrel subdermal implant; female soccer players; young female athletes
MeSH Terms: interventions — etonogestrel; Drug Implants

STUDY DESIGN:
Intervention Model Description: IMPLANON NXT® 68mg:
  Each implant contains 68 mg of etonogestrel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Users of etonogestrel subdermic implant (ESI) (Experimental): 20 female soccer players, under 17 years, who choose subdermic etonogestrel implant (Implanon NXT) as contraceptive . IMPLANON NXT® 68mg (each implant contains 68 mg of etonogestrel) will be the intervention administered.
  Interventions: Device: Implanon NXT® subdermal implant; Drug: Etonogestrel 68mg implant
- Non users of etonogestrel subdermic implant (ESI) (No Intervention): 20 female soccer players without use of any hormonal contraceptive

INTERVENTIONS:
Device: Implanon NXT® subdermal implant — Each implant contains 68 mg of etonogestrel. The release rate is approximately 60-70 mcg/day in the 5th-6th week and reduces to approximately 35-45 mcg/day at the end of the first year; 30-40 mcg/day at the end of the second year and 25-30 mcg/day at the end of the third year.
  It will be evaluation before, 3, 6, 9 and 12 months after implant insertion.Participants' use of the device will be evaluated for one year
  Other Names: Implanon NXT
  Arms: Users of etonogestrel subdermic implant (ESI)
Drug: Etonogestrel 68mg implant — Each implant contains 68 mg of etonogestrel. The release rate is approximately 60-70 mcg/day in the 5th-6th week and reduces to approximately 35-45 mcg/day at the end of the first year; 30-40 mcg/day at the end of the second year and 25-30 mcg/day at the end of the third year.
  It will be evaluation before, 3, 6, 9 and 12 months after implant insertion.Participants' use of the device will be evaluated for one year
  Arms: Users of etonogestrel subdermic implant (ESI)

SUMMARY:
The goal of this clinical trial study is to evaluate the effect of subdermic etonogestrel implant on body composition, sport performance parameters, quantify bleeding patters and quality of life parameters among young female soccer players.

DETAILED DESCRIPTION:
Studies indicate a worsening of performance in young people with excessive menstrual bleeding and menstrual cramps. Hormonal contraception has been used to "manipulate" menstrual symptoms among physically active women, amateur and elite athletes. The use of the etonogestrel subdermal implant (Implanon NXT) would be a good option for young female soccer players. The goal of this study is to evaluate some parameters among young female soccer players under 17 years old during one year, in use of subdermic etonogestrel implant comparing with a non-users subdermic etonogestrel implant

ELIGIBILITY:
Inclusion Criteria:

- sexually active women of childbearing potential, with no contraindications to the use of a progestogen and who agreed to participate in this study.

Exclusion Criteria:

* breastfeeding, irregular vaginal bleeding, increased risk of thromboembolism, ischemic heart disease or other medical conditions

Ages: 16 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Anthropometric Measurements | Clinical, body composition and sport parameters will be evaluation before, 3, 6, 9 and 12 months after implant insertion.
  Weight in kilograms
anthropometric measurements | Will be evaluation before, 3, 6, 9 and 12 months after implant insertion.
  skinfolds in millimeters
anthropometric measurements | Will be evaluation before, 3, 6, 9 and 12 months after implant insertion.
  Height in meters
Body Composition | Will be evaluation before, 3, 6, 9 and 12 months after implant insertion.
  Weight in kilograms and skinfolds in millimeters will be used to measure the athletes' body composition (body composition is used to assess an individual's percentage of body fat and percentage of fat-free mass)
anthropometric measurements | will be evaluated before, 3, 6, 9 and 12 months after implant insertion.
  Weight (in kilograms) and height (in meters) will be used to obtain the BMI (body mass index) (kg/m²)

SECONDARY OUTCOMES:
Sports Performance Parameters | sport parameters will be evaluation before, 3, 6, 9 and 12 months after implant insertion.
  * Kicking Tests : It consists of targets set on a goalkeeper divided into sectors with specific scores, and the numerical values reflect the accuracy of the shot.The goalkeeper is divided into 6 horizontal sectors, with scores assigned to each sector. For example:
  * Lower and central sectors: 2 points.
  * Upper and lateral sectors: 4 points.
  * Shots off goal: 0 points. The player takes 10 shots from within a delimited area (usually the penalty spot).The total points obtained in the 10 kicks are added together.
Sports performance parameters | Will be evaluated before, 3, 6, 9 and 12 months after implant insertion.
  Dribbling test: evaluates ball control and agility, challenging the player to maneuver the ball through obstacle courses in a limited time without losing control.The course is set up with cones spaced alternately in a straight line:
  * Cones positioned every 2 meters, totaling 5 cones on a 10 meter path.
  * The start and finish line is marked. Test Execution
    1. The athlete starts behind the starting line with the ball positioned on the ground.
    2. On command, the athlete dribbles the ball around the cones to the end line, returning to the starting point (round trip).
    3. The test is timed from start to finish. Scoring and Numerical Values
  * Total Time: Performance is recorded in seconds
  * Penalties:
  * Each cone dropped or incorrectly deflected adds 2 seconds to the final time.
  * Losing control of the ball outside the path adds 1 second per occurrence.
  * Evaluation Criteria: Excellent: ≤ 10 sec; Good:10.1 to 12 sec , Regular: 12.1 to 14 sec and Weak > 14

OTHER OUTCOMES:
Bleeding pattern | sport parameters will be evaluation before, 3, 6, 9 and 12 months after implant insertion.
  The bleeding pattern will be classified as favorable or unfavorable:
  Favorable means regular menstrual cycle, between 21 and 35 days, lasting 3 to 7 days and the volume of blood loss does not bother the patient.
  Unfavorable means a cycle lasting less than 21 days, excessive bleeding lasting more than 7 days, intermenstrual bleeding
Quality of life assessment | Quality of life will be evaluated before, 6 and 12 months after implant insertion.
  Quality of life will be measured through the application of the Brief Version in the World Health Organization Quality of Life Brief Version Questionnaire. It is a 26-item self-report questionnaire that assesses quality of life in four domains: physical health, psychological health, social relationships, and environment. Also includes two items that measure overall quality of life and general health.
  The World Health Organization Quality of Life Brief Version scale uses a 5-point Likert scale to score responses to 26 items. The scores are then transformed to a 0-100 scale, with 0 representing the worst possible health status and 100 representing the best

CONTACTS AND LOCATIONS:
Overall Officials: Maíta Poli Araújo, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Department of Gynecology of Federal University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be authorized because the sample is made up of minors and the information collected is confidential. After the study is completed, the results will be duly published in accordance with ethical standards.